CLINICAL TRIAL: NCT04300543
Title: MicroRNA-150 and microRNA-155 as Molecular Biomarkers in Multiple Sclerosis
Brief Title: MicroRNA-150 and microRNA-155 in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamia Ahmed, Administrator, Assiut University
Other Study IDs: MicroRNAs in MS
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: MicroRNA in MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 MS patients: patients with multiple sclerosis
- Group 2 patients with other neurological disorders: patients with inflammatory or non inflammatory neurological diseases other than multiple sclerosis
- Group 3 healthy control: No neurological or immunological disease

SUMMARY:
A study To analyse the expression of circulating miR-150 and miR-155 in serum of MS patients, Evaluate the serum levels of oligoclonal bands, neurofilaments and chitinase-3-like-1 in serum of MS patients, and Investigate the correlation between the measured biomarkers and each other and their correlation with different MS phenotypes , disability status and the patients demographic data.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic neurodegenerative autoimmune disease characterized by infiltration of immune cells into the central nervous system (CNS) with subsequent demyelination, axonal degeneration and neuronal death MS is the most common cause of non traumatic lifelong disability in young adults, affecting women almost three times as often as men

The incidence of MS is increasing worldwide, together with the socioeconomic impact of the disease There is no definite measure or laboratory marker for the diagnosis of MS yet In a patient presenting with an attack, the most important paraclinical test is magnetic resonance imaging (MRI) with intravenous (iv) contrast agent containing gadolinium. This can both present the nature of the lesions (inflammatory and demyelinating characteristics) for differential diagnosis, and the distribution of the lesions within the CNS (evidence of dissemination in time [DIT] and space [DIS] according to the latest McDonald Criteria (2017) Clinical and imaging findings that may be seen in MS, can also be mimicked by some infectious, neoplastic, genetic, metabolic, vascular and other idiopathic inflammatory demyelinating disorders (IIDD) Therefore, to identify MS-related attacks and determine the final diagnosis is vital for the correct treatment choice and longterm disability prevention.

The currently used biomarkers for diagnosing of MS include IgM and IgG antibodies , chemokines, glycoproteins and cell surface markers of inflammation . However, the disease course is very diverse and the heterogenesity in its phenotype not well correlated with biomarkers currently used thus, it is compulsory to identify new specific biomarkers that can help in distinguishing the different MS phenotypes , anticipate the progress of the disease and afford a correlate with the disability status

So, why are biomarkers for MS still arousing interest? Emerging biomarkers, such as circulating miRNAs, display several advantageous features in comparison with previous methods , The possibility to support the results of the clinical diagnosis distinguishing MS subtypes (PPMS, RRMS, etc.) and quantify MS severity , the fact that collecting blood miRNAs and measuring their expression is easy, poorly invasive, and cheap , the robustness of circulating miRNAs which are highly stable, and the accuracy using composite biomarkers rather than a single one.

MicroRNAs (miRNAs) are small non-coding RNA molecule (containing about 22 nucleotides) found in plants, animals and some viruses, that functions in RNA silencing and post-transcriptional regulation of gene expression.

One miRNA can regulate several targets and one target can be regulated by several miRNAs, so miRNAs have multiple biological functions including cell proliferation and differentiation, as well as immune function

The great stability of miRNAs in body fluids, as well as, the sensitive methods for their detection and quantification has led to circulating miRNAs being investigated as biomarkers for various human diseases New evidence has highlighted that miRNA production and trafficking can be dysregulated in both autoimmmune and neurological disorders.

miRNAs are also dysregulated in MS body fluids, including plasma, serum and cerebrospinal fluid.

So more understanding of altered miRNAs expression pattern has enormous potential to be used as diagnostic biomarkers for MS and for monitoring disease progression as well as developing novel therapeutic strategies.

One miRNA with a role in immune function is miR-150, numerous studies suggest that miR-150 regulates maturation and activation of lymphocytes A recent study confirmed that miR-150 controls B cell development by targeting transcription factor c-myb Subsequent studies showed that miR-150 is inversely associated with immunologic functions of activated B and T cells. miR-150 knockout (KO) mice have been shown to enhance T cell-dependent antibody responses and increased steady-state immunoglobulins

Despite considerable data on this molecule, its role in autoimmune disease in particular in multiple sclerosis (MS) is still unknown , miR-150 levels show promising biomarker potential in MS as it can aid in discriminating RRMS from controls Higher levels observed in patients with CIS who converted to MS compared to non converters suggest an involvement in MS progression . So miR-150 may be a novel biomarker of inflammatory active disease with the potential to be used for early diagnosis of MS Another microRNA involved in immune mechanisms is miR-155 which considered a central proinflammatory mediator of CNS It plays a critical role in hematopoietic cell development and tightly regulates innate and adaptive immune responses in response to infection. its dysregulation, more specifically its overexpression, is closely associated with various inflammatory disorders. Although many advances have been made understanding the role of miR-155 in immune cell function and regulation, there are many gaps in understanding its role in non-immune cells. Furthermore, the exact contribution of miR-155 in MS has not been directly explored to understand whether miR-155 is simply a marker for inflammation or whether it plays a predominant role in triggering MS.

Oligoclonal bands are bands of immunoglobulins that are seen when MS patient's blood serum and CSF are analyzed in parallel They are created by immunoglobulin G (IgG) and M (IgM) produced by plasma cells ,they found in nearly all patients with clinically definitive MS. However, OCB are not MS specific and can also occur in other inflammatory CNS diseases . If other diagnoses are excluded though, OCB support the diagnosis of MS. The detection of oligoclonal IgG bands in CSF is associated with a conversion from CIS to MS and can therefore be described as a biomarker for MS prognosis.

Neurofilaments (NF) are neuronal cytoskeletal proteins consisting of a light (NFL), an intermediate (NFM), and a heavy (NFH) chain . They determine the diameter of axons and are involved in axonal transport. If axonal or neuronal damage occurs, NF are released and can be detected in the CSF and blood.

Neurofilaments are emerging as promising new biomarkers for MS, their relative stability and abundance in CNS tissue make them ideal biomarker candidates to monitor ongoing axonal injury and neurodegeneration While these studies are promising, more studies are necessary to determine the sensitivity and specificity of these biomarkers. And a remaining concern regarding neurofilament testing in CSF is the need for repeated LP. So, whether blood levels of neurofilaments sufficiently correlate with disease activity and axonal loss remains to be determined.

Chitinase-3-like-1 Is chitin-binding protein homologous to chitinases, but lacking their capacity for chitin hydrolysis. In MS brain tissue, CHI3L1 (also known as YKL-40) is expressed in astrocytes in white matter plaques and in normal appearing white matter, and is also expressed in microglia in MS lesions. Elevated levels were found in optic neuritis, CIS and MS, So considered as prognostic biomarker for conversion from CIS or optic neuritis to definite MS. But, Its role as a biomarker for disease activity or disease progression is less clear. As its ability to discriminate between SPMS/PPMS and RRMS is not consistent .It also remains unclear whether serum levels of CHI3L1 can provide the same prognostic value as CSF levels

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as MS (clinically and by imaging) according to revised 2017 McDonald Criteria .

Each patient will be subjected to complete medical history uptake including : Age, Sex, age at onset of the disease, phenotype of the disease and its duration, frequency of relapses and remissions , EDSS(The Expanded Disability Status Scale ) is a method of quantifying disability in multiple sclerosis) and MRI findings.

Exclusion Criteria:

* Patients with non neurological autoimmune diseases, malignancy, cardiac and renal diseases that can affect level of miRNAs .

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 140 participants will be enrolled into a study to examine the microRNA and other mentioned biomarkers in their serum, Study population will consist of a total of :80 MS patients recruited among the attendants of out and in patients of neuropsychatric department, 40 with other neurological diseases , 20 healthy control
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
analyse the expression of circulating miR-150 and miR-155 in serum of MS patients | baseline
  to measure the levels of miR-150 and miR-155 in different MS phenotypes
Evaluate the serum levels of oligoclonal bands, neurofilaments and chitinase-3-like-1 in serum of MS patients | baseline
  measure the levels of OCB, NF-L and NF-H , and CHI3L1 in different MS phenotypes

SECONDARY OUTCOMES:
Investigate the correlation between the measured biomarkers and each other and their correlation with different MS phenotypes , disability status and the patients demographic data | baseline
  investigate if the measured biomarkers can distinguish between MS phenotypes, and if they correlate with each other and with the disability status and the patients demographic data

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Eldeek, Ph.D., Study Director — Assiut University; Sally Mohamed, Study Director — Assiut University; Lamia Ahmed, Principal Investigator — Assiut University

REFERENCES:
- [Background] Bergman P, Piket E, Khademi M, James T, Brundin L, Olsson T, Piehl F, Jagodic M. Circulating miR-150 in CSF is a novel candidate biomarker for multiple sclerosis. Neurol Neuroimmunol Neuroinflamm. 2016 Apr 20;3(3):e219. doi: 10.1212/NXI.0000000000000219. eCollection 2016 Jun. PMID 27144214
- [Background] Jagot F, Davoust N. Is It worth Considering Circulating microRNAs in Multiple Sclerosis? Front Immunol. 2016 Apr 5;7:129. doi: 10.3389/fimmu.2016.00129. eCollection 2016. PMID 27092141
- [Background] Chen C, Zhou Y, Wang J, Yan Y, Peng L, Qiu W. Dysregulated MicroRNA Involvement in Multiple Sclerosis by Induction of T Helper 17 Cell Differentiation. Front Immunol. 2018 Jun 4;9:1256. doi: 10.3389/fimmu.2018.01256. eCollection 2018. PMID 29915595
- [Background] Harris VK, Tuddenham JF, Sadiq SA. Biomarkers of multiple sclerosis: current findings. Degener Neurol Neuromuscul Dis. 2017 Jan 12;7:19-29. doi: 10.2147/DNND.S98936. eCollection 2017. PMID 30050375
- [Background] Hu Z, Cui Y, Qiao X, He X, Li F, Luo C, Wang S, Li C, Dai R. Silencing miR-150 Ameliorates Experimental Autoimmune Encephalomyelitis. Front Neurosci. 2018 Jul 10;12:465. doi: 10.3389/fnins.2018.00465. eCollection 2018. PMID 30050402